CLINICAL TRIAL: NCT06146439
Title: Determination of the Factors Causing Treatment Failure in Children Receiving Oxygen Therapy With High-flow Nasal Cannula Due to Moderate and Severe Respiratory Distress
Brief Title: The Factors Causing Treatment Failure in Children Receiving Oxygen Therapy With High-flow Nasal Cannula
Status: Completed | Type: Observational
Sponsor: Dr. Behcet Uz Children's Hospital (Other)
Responsible Party: Principal Investigator, Derşan Onur, Principal Investigator, Dr. Behcet Uz Children's Hospital
Other Study IDs: HFNC failure
Record Dates: First submitted 2023-11-19; First posted 2023-11-24 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: High-flow Nasal Cannula; Respiratory Distress; Treatment Failure
Keywords: Pediatric; HFNC; Respiratory distress; predictor of failure
MeSH Terms: conditions — Dyspnea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Successful: Patients who do not need advanced respiratory support treatments (invasive and noninvasive mechanical ventilation)
- Failure: Patients who need advanced respiratory support treatments (invasive and noninvasive mechanical ventilation)

SUMMARY:
The goal of this observational study is to identify the variables that predict treatment failure in order to identify the patients in which HFNC treatment may fail and not delay the transition to advanced respiratory support treatments in these patients.

The main questions it aims to answer are:

* What factors contribute to the failure of HFNC treatment in these children?
* What is the frequency of HFNC treatment failure in children with moderate and severe respiratory distress? Researchers will compare the group whose HFNC treatment was successful with the group whose HFNC treatment failed to identify factors that cause treatment failure.

DETAILED DESCRIPTION:
Oxygen therapy with a high-flow nasal cannula (HFNC) is a well-tolerated, relatively new, non-invasive alternative ventilation treatment modality. On the other hand, HFNC failure delays advanced respirator supportive treatments, prolongs hospitalization in the intensive care unit, and emergency department, and causes a significant increase in morbidity and mortality with hypoxemia, neurological impairment, and/or hemodynamic instability. The investigators aimed to identify the variables that predict treatment failure in order to identify the patients in which HFNC treatment may fail and not delay the transition to advanced respiratory support treatments in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe respiratory distress
* Oxygen therapy with high-flow nasal cannula

Exclusion Criteria:

* Chronic lung disease (those with CO2 retention or hypoxia in their daily life)
* Cyanotic congenital heart disease
* Craniofacial malformation
* Trauma patients
* Hypotonic patients
* Cases with tracheostomy
* Patients using HFNC therapy for respiratory support after extubation

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: 1 months-18 years Moderate to severe respiratory distress Oxygen therapy with high-flow nasal cannula
Sampling Method: Non-Probability Sample
Enrollment: 201 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
HFNC treatment outcome (failure or success) | 30 days
  Whether advanced respiratory support treatments (invasive and noninvasive mechanical ventilation) are needed

CONTACTS AND LOCATIONS:
Overall Officials: Derşan Onur, Principal Investigator — Dr. Behcet Uz Children's Hospital
Locations (1):
- Dr Behcet Uz Children's Hospital, Izmir, Turkey (Türkiye)

REFERENCES:
- [Background] Er A, Caglar A, Akgul F, Ulusoy E, Citlenbik H, Yilmaz D, Duman M. Early predictors of unresponsiveness to high-flow nasal cannula therapy in a pediatric emergency department. Pediatr Pulmonol. 2018 Jun;53(6):809-815. doi: 10.1002/ppul.23981. Epub 2018 Mar 12. PMID 29528202
- [Background] Liu J, Li D, Luo L, Liu Z, Li X, Qiao L. Analysis of risk factors for the failure of respiratory support with high-flow nasal cannula oxygen therapy in children with acute respiratory dysfunction: A case-control study. Front Pediatr. 2022 Aug 23;10:979944. doi: 10.3389/fped.2022.979944. eCollection 2022. PMID 36081624
- [Background] Sunkonkit K, Kungsuwan S, Seetaboot S, Reungrongrat S. Factors associated with failure of using high flow nasal cannula in children. Clin Respir J. 2022 Nov;16(11):732-739. doi: 10.1111/crj.13533. Epub 2022 Aug 29. PMID 36038361